CLINICAL TRIAL: NCT06289439
Title: Modulation of Sarcopenia in Older Adult Women by Green Tea Extract
Brief Title: Effect of Green Tea Supplementation in Older Adult Women
Acronym: GTAW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Sanidad de Castilla y León (Other); Instituto de Neurociencia de Castillas y Leon (Other)
Responsible Party: Principal Investigator, Diego Fernandez Lazaro, Professor Doctor, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.05.25
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Female; Older Adults; Sarcopenia
Keywords: sarcopenia; green tea; exercise; quality of life; physical performance; health biomarkers
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Tea

STUDY DESIGN:
Intervention Model Description: Parallel group placebo-controlled randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green tea supplementation group (Experimental): 2 capsules for 10 consecutive weeks, distributed in a single daily oral intake with the main meal
  Interventions: Dietary Supplement: Green tea (Camellia sinensis) 1000 mg as extract
- Placebo supplementation group (Placebo Comparator): 2 capsules for 10 consecutive weeks, distributed in a single daily oral intake with the main meal
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Green tea (Camellia sinensis) 1000 mg as extract — Two capsules per day; Each capsule includes Green Tea Leaf (Camellia sinensis) 5000 mg composed of 500 mg of green tea extract and 250 mg of polyphenols (epicatechin (EC), epigallocatechin (EGC), epicatechin gallato (ECG), and epigallocatechin gallato (EGCG))
  Arms: Green tea supplementation group
Other: Placebo — Two capsules per day; Each capsule includes 100-mg maltodextrin capsules were used as a placebo to match the color and texture of the Green tea tablets to ensure blinding.
  Arms: Placebo supplementation group

SUMMARY:
Introduction: One of the consequences of aging is the decrease in physical performance which can affect the quality of life of older people. Although physical exercise is beneficial in improving this problem, older women do not seem to benefit as much as men. In this sense, the use of ergonomic aids by women could compensate for these issues. Thus, green tea has shown beneficial effects on physical performance in athletes through, among others, improving blood flow and vasodilation, mitochondrial respiration, calcium management, glucose and amino acid uptake, lipid oxidation, modulation of muscle damage, antioxidant effect, and anabolic and catabolic hormones, activation of the hypothalamic-pituitary-adrenal axis, etc. Therefore, the deterioration of physical performance and quality of life of green tea.

Objective: To analyze the effect of supplementation with 1 g/day green tea extract (500 mg of polyphenols) for 10 weeks on quality of life values, physical performance (grip strength, walking speed, and resistance), and health biomarkers (biochemical, hematological, and hormonal) in women over 60 years of age who follow a physical training program.

Methods: A total of 20 female volunteers between 60 and 73 years old (age: 65.9±4.58 years, BMI: 25.09±3.24 and body fat percentage: 32.54±6.39) who followed a physical activity adapted to their age and abilities are the members of this study. The volunteers were divided into two groups: placebo (CG; n = 10) and supplemented with 1 g/day of green tea (GI; n = 10). Different physical tests were performed (grip strength, walking speed and resistance) and the quality of life questionnaire (WHOQOL-BREF) was passed and health biomarkers (biochemical, hematological, and hormonal) were analyzed at the beginning (T1) and at the end of the 10 weeks of intervention (T2).

ELIGIBILITY:
Inclusion Criteria:

* Older adult women between 60 and 80 years old, with the ability to carry out a physical activity program adapted to their age and health condition.

Exclusion Criteria:

1. Functional limitation using the Barthel scale (less than 100 = maximum score) and the Lawton-Brody scale (less than 8 = maximum value).
2. Acute/chronic heart failure with NYHA (New York Heart Association) scale >II.
3. Uncontrolled hypertension (>180/100 mm Hg).
4. Uncontrolled orthostatic hypotension.
5. Uncontrolled atrial or ventricular arrhythmias, aortic dissecting aneurysm, severe aortic stenosis, acute endocarditis/pericarditis.
6. Recent acute myocardial infarction (3 to 6 months) or unstable angina.
7. Acute thromboembolic disease.
8. Acute/chronic respiratory failure.
9. Moderate/severe chronic obstructive pulmonary disease (COPD) with Bodex index C or D.
10. Diabetes mellitus with acute decompensation or uncontrolled hypoglycemia.
11. Recent bone fracture (last month).
12. History of dementia (suspected by the MAP environment and diagnosed).
13. Previous supplementation with amino acids or other nutritional compounds to improve physical performance.
14. Any other circumstance that your doctor considers prevents physical activity.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Older adult women
Enrollment: 120 (Estimated)
Dates: Start 2024-03-05 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Creatine kinase (CK) | first day of study and after 30 days of supplementation (end of study)
  CK is an enzyme expressed by various tissues and cell types; markers of muscle damage
Lactate dehydrogenase (LDH) | first day of study and after 30 days of supplementation (end of study)
  LDH is a catalytic enzyme found in many tissues of the body;markers of muscle damage

SECONDARY OUTCOMES:
Myoglobin (Mb) | 1st and 30th days of the trial
  Mb is a muscle heteroprotein
Alanine Aminotransferase (ALT) | 1st and 30th days of the trial
  markers of liver damage
Aspartate Aminotransferase (AST) | 1st and 30th days of the trial
  markers of liver damage
Interleukin 6 (IL-6) | 1st and 30th days of the trial
  inflammatory marker
C-reactive protein (PCR) | 1st and 30th days of the trial
  inflammatory marker
Testosterone | 1st and 30th days of the trial
  hormonal marker
Cortisol | 1st and 30th days of the trial
  hormonal marker
Miostatin (GDF8) | 1st and 30th days of the trial
  growth factor that limits the growth of muscle tissue
advanced oxidation protein products (AOPP) | 1st and 30th days of the trial
  amino acid oxidation marker
lipid peroxidation (LPO) | 1st and 30th days of the trial
  lipid oxidation marker
Oxygen radical absorption (ORAC) | 1st and 30th days of the trial
  antioxidant strength marker
Total antioxidant status (TAS) | 1st and 30th days of the trial
  antioxidant capacity marker
Total antioxidant capacity (TAC) | 1st and 30th days of the trial
  antioxidant capacity marker
Short Physical Performance Battery (SPPB) | 1st and 30th days of the trial
  Test evaluates three aspects of mobility
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | 1st and 30th days of the trial
  a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, University of Valladolid Soria Campus, Soria, Spain